CLINICAL TRIAL: NCT02088385
Title: Pilot Study of a Randomized Controlled Trial Comparing Hemospray Versus the Combined Conventional Technique for Endoscopic Hemostasis of Bleeding Peptic Ulcers
Brief Title: Hemospray Versus the Combined Conventional Technique for Endoscopic Hemostasis of Bleeding Peptic Ulcers : A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Andrew Kwek Boon Eu, Consultant, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/575/E
Record Dates: First submitted 2014-03-13; First posted 2014-03-14 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-07

CONDITIONS: Bleeding Peptic Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemospray (Experimental): Hemospray (TC-325, Cook Medical Inc, Winston-Salem, NC, USA), an adsorptive nanopowder hemostatic agent
  Interventions: Device: Hemospray
- Combined Conventional Technique (Active Comparator): Standard dual therapy with saline adrenaline injection and hemoclip / heater probe application
  Interventions: Device: Combined Conventional Technique

INTERVENTIONS:
Device: Hemospray
  Arms: Hemospray
Device: Combined Conventional Technique
  Arms: Combined Conventional Technique

SUMMARY:
Hemospray (TC-325, Cook Medical Inc, Winston-Salem, NC, USA), a new adsorptive nanopowder hemostatic agent for endoscopic treatment of high-risk bleeding peptic ulcers, provides significant ease of administration compared to the combined conventional technique of saline-adrenaline injection with mechanical clip or heater probe applications. The Hemospray powder is easily applied on ulcers at difficult endoscopic positions and ulcers with fibrotic bases, where the combined conventional technique has limited efficacy. Building up on preliminary work from small single-arm studies, the investigators aim to establish the efficacy and safety of Hemospray in treating bleeding peptic ulcers in comparison with the combined conventional technique. The investigators propose a pilot study to establish our centre's feasibility of performing a prospective, randomized, parallel group trial, which compares the efficacy of Hemospray with the combined conventional technique, in the endoscopic treatment of high-risk bleeding peptic ulcers. Patients with high-risk bleeding peptic ulcers will be treated with Hemospray to determine its initial hemostasis rate (defined as endoscopically verified cessation of bleeding for at least 5 minutes after endoscopic treatment), rebleeding rate (recurrent hemorrhage during a 4-week period following the initial hemostasis) and its safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Peptic ulcer with high-risk stigmata of recent hemorrhage (Forrest class IA, IB, IIA and IIB)

Exclusion Criteria:

* Patients younger than 21 years of age
* Refusal to participate in study
* Contraindicated for endoscopy
* Pregnant or lactating patients
* Bleeding secondary to non-peptic ulcer source
* Patients requiring mechanical ventilation
* Patients with acute coronary syndrome

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kwek, MBBS, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Hemospray: Hemospray (TC-325, Cook Medical Inc, Winston-Salem, NC, USA), an adsorptive nanopowder hemostatic agent
  Hemospray
- Combined Conventional Technique: Standard dual therapy with saline adrenaline injection and hemoclip / heater probe application
  Combined Conventional Technique
Period: Overall Study
Arm/Group | Hemospray | Combined Conventional Technique
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemospray | Combined Conventional Technique | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (18.4) | 72.1 (11.4) | 70 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  Singapore | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Re-bleeding Within 4 Weeks
Description: * drop in hemoglobin of at least 2 g/dl, associated with overt signs of GI bleed (melena, and/or hematemesis)
  * fresh blood hematemesis
  * melena with a hemodynamic instability (pulse rate > 100/min, systolic blood pressure < 90 mm Hg)
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hemospray | Combined Conventional Technique
Number analyzed (Participants) | 10 | 10
Participants | 3 | 1

2. Secondary Outcome: Initial Hemostasis Rate
Description: Endoscopically verified cessation of bleeding for at least 5 minutes after treatment.
Time Frame: Within first endoscopy session
Measure: Count of Participants; unit: Participants
Arm/Group | Hemospray | Combined Conventional Technique
Number analyzed (Participants) | 10 | 10
Participants | 9 | 10

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Hemospray | Combined Conventional Technique
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemospray (N=10) | Combined Conventional Technique (N=10)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — COD pneumonia following surgery for retroperitoneal extension of duodenal ulcer.
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes